CLINICAL TRIAL: NCT04751136
Title: Phase (2) Clinical Trial Studying the Effect of Cerebrolysin on Physical and Mental Functions of Down Syndrome
Brief Title: the Effect of Cerebrolysin on Physical and Mental Functions of Down Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Yahya Wahba, Assistant Professor of Pediatrics and Genetics, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MansouraUCH1
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — cerebrolysin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): infants were given Cerebrolysin®, manufactured by Neuro Pharma Gmbh, in a dose of 0.1 ml / kg body weight once weekly intramuscular injection for 12 month (total of 48 injections).
  Interventions: Drug: cerebrolysin
- Non-intervention Arm (No Intervention): No medication was given

INTERVENTIONS:
Drug: cerebrolysin — Infants of the treatment group were given Cerebrolysin in a dose of 0.1 ml / kg body weight once weekly intramuscular injection for 12 month (total of 48 injections).Each selected infant, in both treatment and control group, was assessed as regard: Socioeconomic status, Nutritional status and feeding practice, assessed for neurocognitive development
  Arms: Intervention Arm

SUMMARY:
Down syndrome is a genetic disorder that causes delay in both physical growth and mental development. It is the most frequently reported chromosomal abnormality and the most common genetic syndrome.

Down syndrome is caused by trisomy of all or part of the genetic material of human chromosome 21. It is now estimated that 94% of individuals with Down syndrome have an extra chromosome 21 as a result of meiotic non-disjunction, or the abnormal segregation of chromosomes during maternal gamete formation and of the remaining 5%, less than 1% is due to somatic mosaicism and the rest is due to chromosome 21 translocations.

The estimated incidence of Down syndrome is between 1 / 1,000 to 1 / 1,100 live births worldwide. In Egypt, the incidence of Down syndrome has been reported to be 1 / 1000 live births.

Down syndrome is characterized by intellectual disability, short stature, distinctive facial characters and a number of co-morbidities including cardiac and digestive anomalies, thyroid problems, and childhood leukemia.

Down syndrome infants will likely experience delays in certain areas and aspects of development. However, they will achieve all of the same milestones as other normal children, just on their own timetable.

According to recent studies, the Down syndrome behavioral phenotype includes relative strengths in some aspects of visuo-spatial processing and social functioning as well as relative deficits in verbal processing. Language has been described as a "major area of deficit" in Down syndrome individuals with particular difficulties manifested in expressive language.

Due to this high incidence of Down syndrome in Egypt and the associated co-morbidities, governmental care directed to this syndrome and other handicapping conditions has increased tremendously in the past few years to the extent that Down syndrome phenotype has become a phobia and many parents and/or physicians referred normal babies for karyotype due to either suspicion of chromosomal anomalies or just for reassurance of their parents.

Although there has been enormous progress in the management of the physical aspects of Down syndrome e.g. repair of heart defects, little advancement has been made to prevent deterioration of cognitive function in these individuals. As a result, the dramatic increase in life expectancy of children with Down syndrome in the past few decades has not been paralleled with concurrent treatment for cognitive disabilities. Therefore, it has remained the most common cause of cognitive dysfunction in children.

The pathogenesis of cognitive deficits and motor disabilities in Down syndrome individuals can be attributed to diminished number and size of neuronal density, progressive neuronal degeneration, impairment of neurogenesis, and reduction in dendrite formation as well as spine density which results in disruption of synaptic function and plasticity. Therefore, many of these individuals develop increasing problems with learning and memory in later life.

Cerebrolysin® is a neurotrophic peptidergic mixture isolated from pig brain. It is produced by standardized enzymatic breakdown of lipid-free porcine brain proteins .

It acts similar to endogenous neurotrophic factors in the form of promoting neuronal sprouting, stimulating neurogenesis, enhancing neuronal plasticity, and improving learning and memory.

Several studies demonstrated that Cerebrolysin® can be used safely in the management of children with any of the following medical conditions: minimal cerebral dysfunction, resistant forms of nocturnal enuresis, neurosensory hypoacusis, attention deficit hyperkinetic disorder, autism and Asperger syndrome.

The overall aim of the study is to assess the effect of Cerebrolysin® on neurocognitive development of infants with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Infants were confirmed to have Down syndrome of non disjunction genotype.
* Age was around 6 month, at time of recruitment.
* Legal guardians accepted to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients having uncontrolled hypothyroidism
* Patients with brain malformations other than the expected in infant with Down syndrome.
* Patients with hearing and / or vision impairments.
* severe congenital heart disease
* Patients having contraindications for the use of Cerebrolysin

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of neurocognitive development | Time frame: 12 month
  We measure neurocognitive development using Bayley Scales of infant and toddler development®, 3rd Edition (BSID -III®) for infants of both groups, after 6 and 12 month of Cerebrolysin® injection. This scale assesses 5 subsets: receptive communication, expressive communication, fine motor, gross motor and cognitive development. Tests are implemented using the child's age (in months) to determine the starting test item for each subtest, and applying the reversal and discontinue rules. Then, the raw score is calculated for each subset as the number of test items that precede the starting item plus the number of items completed by the infant. Finally, test raw scores are recorded on standard record forms. Then, Z scores of scores are calculated according to USA norms. These calculated z scores are used as a standard to compare the rate of development for each subset.

SECONDARY OUTCOMES:
Number of participants with side effects of cerebrolysin | Time frame: 12 month
  We measure side effects that might occur during Cerebrolysin® therapy (one course with total of 48 injections).This is done, with every follow up visit, by physical examination of infants, and history taking from parents and care givers about development of irritability or convulsions during Cerebrolysin® therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sohier Yahia, MD, Study Director — Mansoura University Children Hospital
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valenti D, Braidy N, De Rasmo D, Signorile A, Rossi L, Atanasov AG, Volpicella M, Henrion-Caude A, Nabavi SM, Vacca RA. Mitochondria as pharmacological targets in Down syndrome. Free Radic Biol Med. 2018 Jan;114:69-83. doi: 10.1016/j.freeradbiomed.2017.08.014. Epub 2017 Aug 31. PMID 28838841
- [Background] Baburamani AA, Patkee PA, Arichi T, Rutherford MA. New approaches to studying early brain development in Down syndrome. Dev Med Child Neurol. 2019 Aug;61(8):867-879. doi: 10.1111/dmcn.14260. Epub 2019 May 17. PMID 31102269
- [Background] El-Gilany AH, Yahia S, Shoker M, El-Dahtory F. Cytogenetic and comorbidity profile of Down syndrome in Mansoura University Children's Hospital, Egypt. Indian J Hum Genet. 2011 Sep;17(3):157-63. doi: 10.4103/0971-6866.92092. PMID 22345986
- [Background] Sheets KB, Crissman BG, Feist CD, Sell SL, Johnson LR, Donahue KC, Masser-Frye D, Brookshire GS, Carre AM, Lagrave D, Brasington CK. Practice guidelines for communicating a prenatal or postnatal diagnosis of Down syndrome: recommendations of the national society of genetic counselors. J Genet Couns. 2011 Oct;20(5):432-41. doi: 10.1007/s10897-011-9375-8. Epub 2011 May 27. PMID 21618060
- [Background] Grieco J, Pulsifer M, Seligsohn K, Skotko B, Schwartz A. Down syndrome: Cognitive and behavioral functioning across the lifespan. Am J Med Genet C Semin Med Genet. 2015 Jun;169(2):135-49. doi: 10.1002/ajmg.c.31439. Epub 2015 May 18. PMID 25989505
- [Background] Tsao R, Kindelberger C. Variability of cognitive development in children with Down syndrome: relevance of good reasons for using the cluster procedure. Res Dev Disabil. 2009 May-Jun;30(3):426-32. doi: 10.1016/j.ridd.2008.10.009. Epub 2008 Nov 25. PMID 19036558
- [Background] Weston NM, Sun D. The Potential of Stem Cells in Treatment of Traumatic Brain Injury. Curr Neurol Neurosci Rep. 2018 Jan 25;18(1):1. doi: 10.1007/s11910-018-0812-z. PMID 29372464
- [Background] Muresanu DF, Heiss WD, Hoemberg V, Bajenaru O, Popescu CD, Vester JC, Rahlfs VW, Doppler E, Meier D, Moessler H, Guekht A. Cerebrolysin and Recovery After Stroke (CARS): A Randomized, Placebo-Controlled, Double-Blind, Multicenter Trial. Stroke. 2016 Jan;47(1):151-9. doi: 10.1161/STROKEAHA.115.009416. Epub 2015 Nov 12. PMID 26564102
- [Background] Kim JY, Kim HJ, Choi HS, Park SY, Kim DY. Effects of Cerebrolysin(R) in Patients With Minimally Conscious State After Stroke: An Observational Retrospective Clinical Study. Front Neurol. 2019 Aug 2;10:803. doi: 10.3389/fneur.2019.00803. eCollection 2019. PMID 31428035
- [Background] Krasnoperova MG, Bashina VM, Skvortsov IA, Simashkova NV. [The effect of cerebrolysin on cognitive functions in childhood autism and in Asperger syndrome]. Zh Nevrol Psikhiatr Im S S Korsakova. 2003;103(6):15-8. Russian. PMID 12872620